CLINICAL TRIAL: NCT01701349
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Fosbretabulin Tromethamine (CA4P) in Combination With Paclitaxel and Carboplatin in Anaplastic Thyroid Carcinoma (FACT2)
Brief Title: Fosbretabulin or Placebo in Combination With Carboplatin/Paclitaxel in Anaplastic Thyroid Cancer
Acronym: FACT2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Expected inability to recruit study participants in a reasonable amount of time.
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OX4317s
Record Dates: First submitted 2012-10-02; First posted 2012-10-05 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Anaplastic Thyroid Cancer
Keywords: ATC; Anaplastic Thyroid Cancer; Stage IVC Anaplastic Thyroid Cancer; Thyroid Cancer; Head and Neck Tumors
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms; Head and Neck Neoplasms | interventions — fosbretabulin; Paclitaxel; Carboplatin; combretastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fosbretabulin + paclitaxel + carboplatin (Active Comparator): Six 21 day cycles of:
  Fosbretabulin (60 mg/m2) IV on Day 1, 8, 15 Paclitaxel (200 mg/m2) IV on Day 2 Carboplatin (AUC 6) IV on Day 2
  Interventions: Drug: Fosbretabulin + paclitaxel + carboplatin
- Placebo + paclitaxel + carboplatin (Placebo Comparator): Six 21-day cycles of:
  Placebo (formulated and packages to match fosbretabulin)on Day 1, 8, 15 Paclitaxel (200 mg/m2) IV on Day 2 Carboplatin (AUC6) IV on Day 2
  Interventions: Drug: Placebo + paclitaxel + carboplatin

INTERVENTIONS:
Drug: Fosbretabulin + paclitaxel + carboplatin — Fosbretabulin 200 mg/m2 IV infusion
  Other Names: Fosbretabulin; Combretastatin; Zybrestat; CA4P
  Arms: Fosbretabulin + paclitaxel + carboplatin
Drug: Placebo + paclitaxel + carboplatin — Paclitaxel 200 mg/m2, Carboplatin AUC 6 IV infusion
  Other Names: Paclitaxel; Carboplatin
  Arms: Placebo + paclitaxel + carboplatin

SUMMARY:
This is a multicenter, double-blind, placebo-controlled, randomized study of fosbretabulin given with chemotherapy (paclitaxel and carboplatin) compared to placebo given with chemotherapy (paclitaxel and carboplatin) in subjects with anaplastic thyroid cancer (ATC). The primary objective of the study is to determine overall survival. A maximum of 300 subjects will be recruited from approximately 75 multinational sites of which approximately 35 will be located in the United States.

DETAILED DESCRIPTION:
The Treatment Plan followed for all subjects will consist of:

* A Screening Visit within 14 days before study drug (fosbretabulin or placebo) administration
* A Treatment Phase of 21-day combination treatment (study drug plus chemotherapy) cycles (up to 6 cycles)
* An End of Treatment Phase assessment
* An End of Study Visit occurring 30 days after the last day of study drug administration, as able

After the last clinic visit, all subjects will be followed for survival by monthly phone calls, email, or in-person.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, residual, recurrent or persistent ATC, histologically or cytologically confirmed
* Prior cytotoxic therapeutic regimen as primary therapy for curative intent or prior targeted therapies (TKIs) are eligible (Prior taxane or platinum therapy is allowed)
* Untreated ATC following biopsy, surgery for curative intent, palliation, or after radiation therapy has been considered or administered with or without radiosensitizing chemotherapy
* Disease present on clinical exam (measurable or non-measurable)
* Distant metastases (Stage IVC) only must have histologic confirmation of ATC either from the original primary lesion or a metastatic site
* Neoadjuvant therapy with radiation and either radiosensitizing chemotherapy followed by surgery for curative intent, palliation, or biopsy are eligible if residual or persistent ATC is present
* Subjects with tracheostomy are eligible
* ECOG PS 2 or less
* Adequate bone marrow, renal, and hepatic function, electrolytes WNL for the institution

Exclusion Criteria:

* Disease that is able to be completely resected with negative microscopic margins and without any residual disease in the body
* Active brain metastases, including symptomatic involvement, evidence of cerebral edema by prior CT or MRI, radiographic evidence of brain metastasis since definitive therapy, or continued requirement for corticosteroids for cerebral edema
* History of malignancies other than ACT except prior lower grade thyroid malignancy, curatively treated basal cell carcinoma and in-situ melanoma of the skin, cervical intra-epithelial neoplasia,localized prostate cancer, in-situ carcinoma of the breast
* Known intolerance or hypersensitivity to fosbretabulin, paclitaxel, carboplatin or any of their components
* Receiving concurrent investigational therapy or have received investigational therapy for any indication within 28 days of the first scheduled day of dosing
* Grade 3 or greater peripheral neuropathy
* History of prior cerebrovascular event,including transient ischemic attack within the past 6 months
* Uncontrolled hypertension defined as blood pressure >150/100 mm Hg despite medication
* Symptomatic vascular disease (e.g. intermittent claudication)
* History of unstable angina pectoris pattern, myocardial infarction (including non-Q wave) within the past 6 months, or NYHA Class III or IV congestive heart failure
* History of torsade de pointes, ventricular tachycardia, ventricular fibrillation or congenital long QT syndrome.
* Pathologic bradycardia (<60 b/m or heart block(excluding 1st degree block, consisting of PR interval prolongation only)
* ECG findings of clinically significant ventricular arrhythmia, new ST segment elevation or depression, or new Q wave on ECG (PVCs are not excluded).
* QTc interval 480 ms or more
* Requirement of concurrent treatment with any drugs know to prolong the QTc interval, including anti-arrhythmic medications
* Potassium and/or magnesium concentrations below normal range for the reference laboratory
* History of solid organ or bone marrow transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Maximun length of study for each subject is 2 years from date of randomization

SECONDARY OUTCOMES:
Number of adverse events of the combination of fosbretabulin + paclitaxel + carboplatin | Maximun length of study for each subject is 2 years from date of randomization
Number of participants with 1-year survival | Maximun length of study for each subject is 2 years from date of randomization

OTHER OUTCOMES:
Determine the proportion of subjects with measurable disease who have objective tumor response, by treatment | Maximun length of study for each subject is 2 years from date of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Brose, MD, PhD, Principal Investigator — University of Pennsylvania, Philadelphia, PA 19104; Julie A Sosa, MD, Principal Investigator — Yale University, New Haven, CT 06520; Lisa Licitra, MD, Principal Investigator — Instituto Nazionale Per Lo Studio E La Cura Dei Tumori, Milan, Italy

REFERENCES:
- See also: Thyroid Cancer Survivors' Association, Inc. — http://thyca.org